CLINICAL TRIAL: NCT03835871
Title: A Randomized, Parallel Group, Multicenter, Double -Blind, Double-dummy, Placebo-controlled Phase 3 Study With Beclomethasone Dipropionate HFA at 100 μg, 200 μg and 400 μg Daily Doses Compared to Placebo in Mild or Moderate Persistent Asthma
Brief Title: Beclomethasone Dipropionate HFA in Adult and Adolescent Subjects With Mild to Moderate Persistent Asthma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Adamis Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-1000-03
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double -blind, double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 400 µg per day Beclomethasone (Experimental): Intervention: Drug: Beclomethasone 400 µg per day Daily dose of Beclomethasone 400 µg 2 inhalations 100 μg ex-valve 2 times a day for 12 weeks
  Interventions: Drug: 400 µg per day Beclomethasone
- 200 µg per day Beclomethasone (Experimental): Intervention: Drug: Beclomethasone 200 µg per day Daily dose of Beclomethasone 200 µg 1 inhalation 100 μg ex-valve 2 times a day for 12 weeks Intervention: Drug: Placebo 1 inhalation 2 times a day for 12 weeks
  Interventions: Drug: Placebo; Drug: 200 µg per day Beclomethasone
- 100 µg per day Beclomethasone (Experimental): Intervention: Drug: Beclomethasone 100 µg per day Daily dose of Beclomethasone 100 µg 1 inhalation 50 μg ex-valve 2 times a day for 12 weeks Intervention: Drug: Placebo 1 inhalation 2 times a day for 12 weeks
  Interventions: Drug: Placebo; Drug: 100 µg per day Beclomethasone
- placebo (Placebo Comparator): Intervention: Drug: placebo 2 inhalations 2 times a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Intervention: Drug: placebo
  Other Names: placebo for Beclomethasone Dipropionate HFA
  Arms: 100 µg per day Beclomethasone; 200 µg per day Beclomethasone; placebo
Drug: 400 µg per day Beclomethasone — Intervention: Drug: Beclomethasone 400 µg HFA per day
  Other Names: Beclomethasone Dipropionate HFA
  Arms: 400 µg per day Beclomethasone
Drug: 200 µg per day Beclomethasone — Intervention: Drug: Beclomethasone 200 µg HFA per day
  Other Names: Beclomethasone Dipropionate HFA
  Arms: 200 µg per day Beclomethasone
Drug: 100 µg per day Beclomethasone — Intervention: Drug: Beclomethasone 100 µg HFA per day
  Other Names: Beclomethasone Dipropionate HFA
  Arms: 100 µg per day Beclomethasone

SUMMARY:
Approximately 480 (120 per group) would need to complete the 12 weeks of treatments.

DETAILED DESCRIPTION:
This is four arm study. Approximately 480 (120 per group) would need to complete the 12 weeks of treatments.In order to achieve that number of subjects, approximately 700 subjects will be screened randomized into the study.

A screening visit (Visit 1) will be followed by at least 2 weeks (14 days) placebo Run-in Period during which asthma subjects will wash out their daily inhaled corticosteroid and other medications and be assessed for compliance.

Study treatment period will be for a duration of 12 weeks with visits: Visit 2- Baseline Day 1, Visit 3 Day 21 (± 2 days), Visit 4 Day 42 (± 2 days), Visit 5 Day 63 (± 2 days), and Visit 6 Day 84 days (± 2 days).

Rescue Therapy: Short-acting beta agonists, Albuterol 90 μg/actuation.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects (between ≥ 12 and ≤ 80 years old). Females may be of either childbearing or non-childbearing potential. All females of childbearing potential must be either abstinent from sexual intercourse or using adequate contraception and must also have a negative pregnancy test. Pregnant or nursing females or females intending to become pregnant during the course of the study must be excluded from the study.
2. The subject has mild to moderate asthma as defined by the National Asthma Education a Prevention Program (NAEPP ERP-3 ), at least 12 weeks prior to screening.
3. Pre-bronchodilator forced expiratory volume in 1 second (FEV1) on the screening visit and on the baseline visit is > 60% of the predicted value of predicted values according to age, height, race and sex using The global lung function 2012 equations: Report of the Global Lung Function Initiative (GLI), following abstinence from short-acting β-agonists for a minimum of 6 hours and withholding restricted medications prior to the visits. At Visit 2 the baseline FEV1 and the predicted FEV1 value would be the mean of 2 pre-dose FEV1 measurements taken 30 minutes apart (-30 min and 0).
4. The subject has demonstrated at least 12% reversibility of FEV1 at either the screening or baseline visit within 30 minutes after 4 inhalations (total of 360 μg) of albuterol (pMDI). [Note: Subjects who fail to demonstrate the required reversibility at the Screening Visit (Visit 1) are eligible to enter the Run-in Period and repeat the testing at the End of Run-in Period/Baseline (Visit 2)].
5. If the subject in on inhaled corticosteroids the subject must be on a stable dose of daily-inhaled corticosteroid (ICS), at least 80 μg/day of beclomethasone dipropionate or equivalent for a minimum of 4 weeks before screening visit
6. Currently nonsmoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and had ≤ 10 pack years of historical use.
7. A body mass index between 18-35 kg/m2, inclusive.
8. Willingness to give their written informed consent/assent to participate in the study.
9. Subjects must be able to perform acceptable and repeatable spirometry, Peak Flow Meter (twice a day measurements), keep a diary record and to use the inhalation devices as assessed at Screening and Baseline by the study staff.
10. Ability to understand and comply with the protocol requirements, instructions and protocol stated restrictions.

NOTE: At the end of the placebo Run-in period the subject will be stratified into two categories:

* Corticosteroid naïve subjects (Not have taken inhaled corticosteroids (ICSs) at least 3 months prior to screening or systemic corticosteroids at least 6 months before screening)
* Prior corticosteroid users

Exclusion criteria

1. Incidence of asthma exacerbations per NAEPP ERP-3(1) (Appendix IV) within the last 3 months.
2. Respiratory diseases other than asthma or allergic rhinitis.
3. Uncontrolled asthma defined as having 3 - 4 of the following symptoms: a) Daytime asthma symptoms (> twice/week) b) Night waking due to asthma c) Reliever needed for symptoms more than twice a week (excluding reliever taken before exercise) d) Any activity limitation due to asthma per GINA, Chapter 2, Box 2-2, page 29.
4. Life threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia; respiratory arrest or hypoxic seizures, asthma related syncopal episode(s) within the previous 10 years.
5. The known presence or history of tuberculosis infection of the respiratory tract; untreated systemic fungal, bacterial, parasitic or viral infections; or ocular herpes simplex.
6. The presence or history of a clinically significant medical condition, other than asthma including laboratory result abnormalities that in the opinion of the investigator would put the subject at risk through study participation or would affect the study analyses if the disease exacerbated during the study. Following conditions should be considered carefully: congestive heart failure, recent myocardial infraction, uncontrolled hypertension, cardiac arrhythmias and diabetes mellitus, epilepsy, glaucoma, cataract, uncontrolled hypothyroidism, liver failure, severe osteoporosis, peptic ulceration and renal impairment.
7. Hospitalization for asthma or a respiratory condition in the last 12 months.
8. Need for oral steroids and/or antibiotics for lung disease in last 3 months.
9. Current or recent respiratory infection or current oral candida infection.
10. Participation in another clinical trial or study within 1 month or at least 5 half-lives (whichever is longer) preceding the first dose of trial medication. Previous participation in this study.
11. Use of any of the following excluded respiratory medications within the indicated time frame prior to screening and throughout the study:

    1. Anti-IgE antibody (e.g. Xolair) and depot corticosteroids 3 months
    2. Systemic (I.V., I.M., oral) corticosteroids 3 months
    3. Inhaled corticosteroids Stop at screening
    4. Long-acting anti-muscarinics (e.g., tiotropium) 48 hours
    5. Short-acting anti-muscarinics (e.g., ipratropium) 24 hours
    6. LABA (e.g., salmeterol, formoterol,etc.) 12 hours
    7. Short-acting β2-adrenergic agonists (SABA), except for study rescue medication (albuterol) 6 hours
    8. Oral β2-adrenergic agonists 1 month
    9. Topical dermatologic corticosteroids of intermediate to high potency such as fluticasone propionate, mometasone furoate 14 days
    10. Oral or nasal antihistamines unless on a stable dose for 30 days prior screening.
    11. Immunologically active biologic medications such as anti-TNFα (tumor necrosis factor) 3 months
    12. Immunosuppressive therapy such as methotrexate, gold, Azathioprine 1 month
    13. Immunotherapy initiation within 3 months or change in dose within 1 month
    14. Over-the-counter bronchodilators 2 weeks
    15. Marijuana 1 month
    16. Inhaled nicotine such as e-cigarettes 1 day
12. Use of the following medications 30 days before screening:

    1. Non-cardio selective β-blockers (e.g. propranolol, nadolol, carvedilol, labetalol, sotalol)
    2. Digitalis
    3. Thiazide diuretics
    4. Oral decongestants
    5. Cytochrome P450 3A4 enzyme inhibitors
    6. Benzodiazepines
    7. Cyclic antidepressants
    8. Monoamine oxidase inhibitors
    9. Diazoxide
    10. Ketoconazole, itraconazole
    11. Phenytoin
    12. Rifampicin
    13. Mifepristone
13. Known hypersensitivity to any corticosteroid or any of the excipients in the study drug or rescue medication formulation.
14. Evidence (as assessed by the Investigator using good clinical judgment) of alcohol or drug abuse or dependency at the time of screening, for the 6 months prior to screening.
15. Live in the same household as currently enrolled subject.
16. Any other reason which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Mean Change from baseline trough (pre-dose and pre-rescue) FEV1 percent predicted at week 12 | 12 weeks
  Mean Change from baseline trough (pre-dose and pre-rescue) FEV1 percent predicted at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Carlo, Study Chair — CEO